CLINICAL TRIAL: NCT06244017
Title: Comparisons Between Electroencephalographic Spectrogram-guided and Bispectral Index-guided Multimodal General Anesthesia During Craniotomy- a Randomized Controlled Trial
Brief Title: EEG Spectrogram-guided vs. Index-guided Anesthesia for Craniotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202312067DINA
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Craniotomy
MeSH Terms: interventions — Consciousness Monitors

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EEG Spectrogram-guided (Experimental): The general anesthesia administration is guided by using the EEG spectrogram in this group. Other perioperative care protocols are the same between the two study group.
  Interventions: Device: EEG spectrogram
- Bispectral index-guided (Active Comparator): The general anesthesia administration is guided by using the processed EEG index, namely the bispectral index (BIS) in this group. Other perioperative care protocols are the same between the two study group.
  Interventions: Device: Bispectral index

INTERVENTIONS:
Device: EEG spectrogram — In the experimental group, the general anesthesia is guided by using the EEG spectrogram.
  Arms: EEG Spectrogram-guided
Device: Bispectral index — In the control group, the general anesthesia is guided by using the bispectral index
  Arms: Bispectral index-guided

SUMMARY:
In this trial, investigators aimed to compared the clinical effects between the electroencephalographic (EEG) spetrogram-guided and processed EEG index-guided multimodal general anesthesia using the combination of propofol, dexmedetomidine, remifentnil and the scalp block in patients undergoing elective craniotomy.

DETAILED DESCRIPTION:
The multimodal general anesthesia involved the administration of combinations of antinociceptive agents and hypnotics using electroencephalographic (EEG) based monitors to achieve a balanced state of anesthesia. Traditionally, the adjustment of general anesthesia drugs has been done using instruments like the Bispectral Index (BIS), which converts frontal lobe EEG signals into a numerical range of 0-100. This allows anesthesiologists to assess drug dosage and depth of anesthesia. However, numerical conversion may not accurately reflect individual variations and cannot precisely calculate drug concentrations in the case of multiple drug combinations.

For instance, dexmedetomidine (DEX) is currently one of the most commonly used drugs in multimodal generagal anesthesia.Because each anesthetic produces distinct brain states that are readily visible in an EEG density spectral array (DSA) and can be easily interpreted by anesthesiologists, anesthetic titration based on an EEG DSA may provide additional information for anesthetic depth monitoring and may avoid the conventional 'one-index-fits-all' approach, which often ignores the influence of anesthetic drug combination. Theoretically, the anesthetic exposure in cases that involve the coadministration of dexmedetomidine can be more precise through the use of an EEG DSA than the use of BIS value. In accordant to this context, investigators have changed our institutional anesthetic propofol from BIS guidance to the DSA guidance and based on the retrospective analysis, investigators further observed the profound anesthetic-sparing effects and potential postoperative benefits of EEG DSA-guided anesthesia comparing to the BIS-guided anesthesia (doi: 10.4097/kja.23118). Therefore, further prospective randomized controlled is warranted to shape the real clinical benefits of DSA-guided multimodal general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective craniotomy

Exclusion Criteria:

* revision surgery
* heart failure
* liver cirrhosis > Child B class
* chronic obstructive pulmonary disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Intraoperative anesthetic dose | 4-6 hours
  We aim to compare the intraoperative propofol consumptions between the two study groups

SECONDARY OUTCOMES:
Postoperative neurological complication incidence | During the hospital stays; approximately 7-10 days
  We aim to compare the postoperative neurological complication incidence between the two study groups

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yu Wu, Principal Investigator — National Taiwan University Hospital Hsinchu Branch
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan